CLINICAL TRIAL: NCT00967408
Title: Effects on Clinical and Functional Outcome of Escitalopram in Adult Stroke
Brief Title: Effects on Clinical and Functional Outcome of Escitalopram in Adult Stroke Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Stefano Carda, MD, Physical medicine & Rehabilitation Dpt. AOU Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49CE 8/08
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Stroke
Keywords: Stroke; Antidepressive Agents,Second-Generation; Treatment Outcome; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation + Escitalopram (Experimental): Rehabilitative treatment + Oral Escitalopram 5 mg/day for the first week, 10 mg/day from second to fourth week and 20 mg/day until 6th month.
  Interventions: Drug: Escitalopram; Other: Rehabilitative treatment
- Rehabilitation + Placebo (Placebo Comparator): Rehabilitative treatment + Non active Placebo tablets for 6 months
  Interventions: Drug: Placebo; Other: Rehabilitative treatment

INTERVENTIONS:
Drug: Escitalopram — Rehabilitative treatment + Oral Escitalopram 5 mg/day for the first week, 10 mg/day from second to fourth week and 20 mg/day until 6th month.
  Other Names: ATC N06AB10
  Arms: Rehabilitation + Escitalopram
Drug: Placebo — Rehabilitative treatment + oral inactive placebo for 6 months
  Arms: Rehabilitation + Placebo
Other: Rehabilitative treatment — Rehabilitative treatment

SUMMARY:
Rehabilitative treatment in stroke survivors has shown to be effective in improving functional outcome and reducing dependency. Plasticity of the central nervous system, along with coping strategies and adaptations, seems to play a key role in functional recovery. Some data support the hypothesis that drug which improve dopaminergic, serotoninergic and noradrenergic transmission in the central nervous system could improve recovery in stroke patients. In this population, antidepressants as selective serotonin reuptake inhibitors (SSRI) are associated to better outcomes, as evidenced by small clinical trials. However, since depression is a common consequence of stroke, observed improvements could be biased by the action of these drugs on depressive symptoms, thus improving participation in rehabilitative treatment.

The hypothesis of this study is that SSRI could improve functional outcome in stroke survivors not only because of their action on depressive symptoms, but mainly because of a direct effect on neural repair and neuronal growth.

The aim of the study is to evaluate the effect of a SSRI, escitalopram, on functional outcome of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* age > 18 years
* first ischaemic and haemorrhagic stroke

Exclusion Criteria:

* unstable medical conditions
* unable to understand study aims and procedures
* severe aphasia
* other progressive neurological disease
* previous or concomitant psychiatric illness
* patients not willing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure | Enrollment, 2 and 6 months

SECONDARY OUTCOMES:
Mini-mental state examination (MMSE) | Enrollment, 2 and 6 months
Trunk Control Test | Enrollment, 2 and 6 months
Canadian Stroke Scale | Enrollment, 2 and 6 months
Motricity Index | Enrollment, 2 and 6 months
Token test | Enrollment, 2 and 6 months
The Bells Test | Enrollment, 2 and 6 months
Stroop Test | Enrollment, 2 and 6 months
Wisconsin Card Sorting test | Enrollment, 2 and 6 months
Verbal Fluency | Enrollment, 2 and 6 months
Raven's Matrices Test | Enrollment, 2 and 6 months
Trail Making A-B Test | Enrollment, 2 and 6 months
Center for Epidemiological Studies Depression Scale | Enrollment, 2 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Physical medicine & rehabilitation Dept AOU Maggiore della Carità, Novara, Italy